CLINICAL TRIAL: NCT04948255
Title: Work-Related Stress Amongst a Primary Care Workforce in Greater Manchester, United Kingdom Before and During the Covid-19 Pandemic
Brief Title: Measuring Work-Related Stress in Primary Care in the Covid-19 Pandemic
Acronym: WRS
Status: Completed | Type: Observational
Sponsor: Dr. Faizan Awan (Other)
Responsible Party: Sponsor-Investigator, Dr. Faizan Awan, General Practitioner, The Gill Medical Centre
Organization: The Gill Medical Centre (Other)
Other Study IDs: 302893
Record Dates: First submitted 2021-06-29; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Occupational Stress; Covid19
Keywords: Pandemics; Primary health care
MeSH Terms: conditions — Occupational Stress; COVID-19 | interventions — Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare Workers at the Gill Medical Centre: Clinical and non-clinical staff at the Gill Medical Centre will complete a validated stress questionnaire during the Covid-19 pandemic. A baseline was established in May, 2019.
  Interventions: Other: Health and Safety Executive's (HSE) Management Standards Indicator Tool (MSIT) to measure work-related stress

INTERVENTIONS:
Other: Health and Safety Executive's (HSE) Management Standards Indicator Tool (MSIT) to measure work-related stress — Questionnaire

SUMMARY:
This prospective cohort study was designed to assess WRS amongst clinical and non-clinical staff in a primary healthcare setting using a validated tool with a view to developing an evidence base to form a historical and comparative record during the Covid-19 pandemic.

DETAILED DESCRIPTION:
Work-related stress (WRS) is the second most common cause of occupational ill health in the United Kingdom. Studies suggest that during the Covid-19 pandemic, an increased prevalence of stress-related disorders was reported amongst healthcare workers. WRS can be assessed using the Health and Safety Executive's (HSE) Management Standards Indicator Tool (MSIT) and is used to compare changes to WRS across six domains over time. Lower scores in domains indicate higher WRS experienced by workers. Increases in the score in subsequent assessments indicate improvements to WRS. The MSIT was distributed to 23 primary care clinical and non-clinical staff in a medical centre in Greater Manchester, United Kingdom in March, 2019. 18 responses were received from 23 staff (78% response rate), establishing a baseline. In May, 2020, the authors decided to reanalyse the effect of the Covid-19 pandemic on WRS upon the same population. The MSIT was redistributed in March 2021, with 14 responses from 20 staff (70% response rate). Microsoft Excel's data analysis was applied to the results. WRS across the practice increased by 7% in demands, 4% in control and 2% in role domains and improved by 3% in support, 3% in relationships and 2% in change domains. The results are in keeping with the global picture of evolving WRS amongst healthcare staff during the pandemic. Monitoring and addressing WRS regularly helps maintain system-wide resilience when faced with unexpected or unprecedented change. Comparing these results with WRS in other healthcare systems would be a useful next step.

ELIGIBILITY:
Inclusion Criteria:

* Primary healthcare staff working at the Gill Medical Centre for at least two months prior to assessment.

Exclusion Criteria:

* Any staff member employed for less than two months, those who were off work due to non- stress related long-term leave or incomplete submissions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult health professionals and administration staff
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Measurement of stress across the workforce | 24 months
  Work-related stress (WRS) is measured using the Management Standards Indicator Tool (MSIT) on a Likert scale of 1-5 with a higher number indicating less WRS. A measurement is made at baseline and during the Covid-19 pandemic.

SECONDARY OUTCOMES:
Measurement of stress by type of role | 24 months
  WRS measured using MSIT across three different primary healthcare roles - doctors, other clinicians and administrators - at baseline from 2019 and during the Covid-19 pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Ashleigh Ward, MBChB, Principal Investigator — Salford Royal Hospital
Locations (1):
- The Gill Medical Centre, Salford, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Sharing of collected data with researchers using the same tool to assess work-related stress.
Supporting Information: SAP, CSR
Time Frame: Data available now 29/06/2021 to 29/06/2031.
Access Criteria: E-mail: faizan@doctors.org.uk with name, contact details and study purpose.